CLINICAL TRIAL: NCT07283705
Title: A Phase II Study Evaluating BMS-986504 in MTAP-deleted Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0804; NCI-2025-09221 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-12-11; First posted 2025-12-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Phase 2 Study; BMS-986504; MTAP-deleted Pancreatic Cancer
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Will receive a combination of BMS-986504, gemcitabine, and nab-paclitaxel for 4 treatment cycles.
  Interventions: Drug: BMS-986504; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Cohort 2 (Experimental): Will receive a combination of BMS-986504, gemcitabine, and nab-paclitaxel for 4-6 months, followed by Maintenance Therapy with BMS-986504 by itself for as long as the disease does not get worse.
  Interventions: Drug: BMS-986504; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Cohort 3 (Experimental): Will receive a combination of BMS-986504, and the combination treatment mFOLFIRINOX (oxaliplatin, irinotecan, and 5-fluorouracil) for 4-6 months.
  Interventions: Drug: BMS-986504; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: BMS-986504 — Given by po
Drug: Gemcitabine — Given by IV
  Arms: Cohort 1; Cohort 2
Drug: Nab-paclitaxel — Given by IV
  Arms: Cohort 1; Cohort 2
Drug: mFOLFIRINOX — Given by iv
  Arms: Cohort 3

SUMMARY:
To find out if the combination of BMS-986504 plus neoadjuvant/adjuvant chemotherapy and surgery (Cohort 1) or BMS-986504 plus standard of care chemotherapy (Cohorts 2 and 3) can help to control pancreatic cancer.

DETAILED DESCRIPTION:
Primary Objectives

* Cohort 1: To evaluate the safety and tolerability of BMS-986504 in combination with neoadjuvant/adjuvant chemotherapy and as maintenance therapy in participants with resectable/borderline resectable PDAC. Major pathological response (MPR) and incidence, severity and duration of pre- and post-operative complications (e.g. delay of surgery, inability to get surgery, type and rate of postoperative complications [like pancreatic fistula], rate of resection for borderline participants) will be evaluated.
* Cohorts 2 and 3: To evaluate the safety, tolerability and efficacy of BMS-986504 in concomitant with SOC chemo and as maintenance therapy. Efficacy will be evaluated as disease control (PFS) at 6 months in participants with locally advanced (Cohort 2) and metastatic (Cohort 3) PDAC.

Secondary Objectives

• To evaluate 6-month overall response rate (ORR) and disease control rate (DCR) for Cohorts 1,2 and 3

ELIGIBILITY:
Eligibility Criteria

* Age ≥18 years.
* Homozygous MTAP deletion detected by NGS. Test can be performed on an archival tissue collected within 6 months from study enrollment and on blood samples.
* ECOG performance status 0-1.
* Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC)
* Adequate organ and marrow function as defined below

  * Hemoglobin ≥9.0 g/dL with no packed red blood cell transfusions in the past 7 days.
  * Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L.
  * Platelet count ≥100 x 10⁹/L with no platelet transfusions in the past 7 days.
  * Total bilirubin ≤1.5 x institutional upper limit of normal (ULN).
  * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional ULN value unless liver metastases are present, in which case ≤5 x ULN.
* Calculated creatinine clearance ≥50 mL/min (using Cockroft-Gault formula or 24-hour urine collection).
* Participants are allowed to have received 1 month of GA (cohort 1 and 2) and mFolfirinox (cohort 3) in consideration of the aggressive nature of PDAC and the time required for to test MTAP-deficiency
* Agree to follow the study protocol, including treatment, scheduled visits, and examinations, for the duration of the study.
* Ability to understand and the willingness to sign a written informed consent document.

  1 Female (as assigned at birth) participants
* Women of child-bearing potential (WOCBP) include all female participants, between the onset of menses and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114): :

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* WOCBP must agree to use a combination of a hormonal and a non-hormonal contraceptive method or a non-hormonal method alone that is highly effective (with a failure rate of < 1% per year) during the intervention period and for at least 9 months after the last dose of study intervention, or according to approved local product label requirements for individual chemotherapy agents, whichever is longer.

  * WOCBP are not permitted to use hormonal contraceptive methods alone as a highly effective method of contraception and must use an additional non-hormonal highly effective method of contraception.
  * WOCBP participants must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction for the same period. Participants should be advised to seek advice about egg donation and cryopreservation of germ cells before treatment.
  * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, and Implantable or injectable contraceptives. . Not engaging in sexual activity for the entire period of risk associated with the study intervention is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

    2 Male (as assigned at birth) participants
* Male (as assigned at birth) participants will be required to always use a latex or other synthetic condom during any sexual activity (eg, vaginal, anal, oral) with WOCBP, even if the participant has undergone a successful vasectomy or if the partner is pregnant or breastfeeding. Male (as assigned at birth) participants should continue to use a condom during the intervention period and for at least 6 months after the last dose of study intervention, or according to approved local product label requirements for individual chemotherapy agents, whichever is longer.
* Male (as assigned at birth) participants with a pregnant or breastfeeding partner must agree to remain abstinent from sexual activity or use a male condom during any sexual activity (eg, vaginal, anal, oral), even if the participant has undergone a successful vasectomy, during the intervention period and for at least 6 months after the last dose of study intervention or according to approved local product label requirements for individual chemotherapy agents, whichever is longer.
* Male (as assigned at birth) participants must refrain from donating sperm during the intervention period and for at least 6 months after the last dose of study intervention, or according to approved local product label requirements for individual chemotherapy agents, whichever is longer. Participants should be advised to seek advice about sperm donation and cryopreservation of germ cells before treatment.
* WOCBP partners of male (as assigned at birth) participants should be advised to use a highly effective method of contraception during the intervention period and for at least 6 months after the last dose of study intervention, or according to approved local product label requirements for individual chemotherapy agents, whichever is longer, for the male participant.

Cohort 1 specific criteria:

* Resectable or borderline resectable pancreatic adenocarcinoma per NCCN version 3.202432 that have not received any neoadjuvant treatment

  o Resectable PDAC will be defined as the tumor with:
* No arterial tumor contact (celiac axis [CA], superior mesenteric artery [SMA], or common hepatic artery [CHA])
* No tumor contact with the superior mesenteric vein (SMV) or portal vein (PV) or ≤180° contact without vein contour irregularity.
* Borderline PDAC will be defined as the tumor with:

  o For tumors of the pancreatic head/uncinate process:
* Solid tumor contact with CHA without extension to CA or hepatic artery bifurcation, allowing for safe and complete resection and reconstruction.
* Solid tumor contact with the SMA of ≤180°.
* Solid tumor contact with variant arterial anatomy (eg, accessory right hepatic artery, replaced right hepatic artery, replaced CHA, and the origin of replaced or accessory artery) and the presence and degree of tumor contact should be noted if present, as it may affect surgical planning.
* Solid tumor contact with the SMV or PV of >180°, contact of ≤180° with contour irregularity of the vein or thrombosis of the vein but with suitable vessel proximal and distal to the site of involvement, allowing for safe and complete resection and vein reconstruction.
* Solid tumor contact with the inferior vena cava (IVC).

  o For tumors of the pancreatic body/tail:
* Solid tumor contact with the CA of ≤180°

Cohort 2 specific criteria:

* Locally advanced, unresectable pancreatic cancer per NCCN version 3.202432

  o For tumors of the head/uncinate process:
* Solid tumor contact >180° with the SMA or CA
* Unreconstructible SMV/PV due to tumor involvement or occlusion (can be due to tumor or bland thrombus).

  o For tumors of the pancreatic body/tail:
* Solid tumor contact of >180° with the SMA or CA.
* Solid tumor contact with the CA and aortic involvement.
* No prior treatment with the exception of one month of chemotherapy with GA without progression of disease

Cohort 3 specific criteria:

* Metastatic pancreatic adenocarcinoma.
* No prior treatment, except one month of chemotherapy with mFOLFIRINOX without progression of disease.

Exclusion Criteria

* Prior treatment with PRMT5 and MAT2A inhibitors.
* Exposure to an investigational agent within 30 days or 5 half-lives (whichever is longer) prior to trial enrolment is not permitted.
* Participants with other primary cancers are excluded, except for adequately treated nonmelanoma skin cancer, prostate cancer post-resection with undetectable PSA, in-situ cervical cancer, ductal carcinoma in situ (DCIS) of the breast, Stage 1 Grade 1 endometrial carcinoma, or solid tumors (including lymphomas without bone marrow involvement) curatively treated with no evidence of disease for ≥2 years prior to study entry.
* Major surgery within 2 weeks of starting treatment is not permitted. Participants must have recovered from the effects of any major surgery.
* Significant third-space fluid retention (e.g., ascites or peritoneal effusion) that requires drainage within 1 month prior to randomization.
* Cardiac abnormalities including:

  * Left ventricular ejection fraction < 50%
  * History of prolonged QTc, or QT interval corrected for heart rate using Fridericia's formula (QTcF) prolongation > 480 msec, except for right bundle branch block
  * Uncontrolled/symptomatic or significant cardiovascular conditions within 6 months prior to enrollment, including but not limited to any of the following:
* Cardiac angioplasty or stenting, myocardial infarction, stroke/transient ischemic attack, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, New York Heart Association (NYHA) class III-IV congestive heart failure, pericarditis, myocarditis, atrial fibrillation or other arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or Torsade's de pointes)
* Ongoing need for a medication with a known risk of Torsade's de Pointes or known as a strong inhibitor or strong inducer of CYP3A4 and/or P-glycoprotein or a proton-pump inhibitor that cannot be switched to alternative treatment prior to study entry. The following drug interaction databases and other literature can be utilized to determine the CYP3A4/Pgp inhibitors and inducers:

  * https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-anddruginteractions- table-substrates-inhibitors-and-inducers.
  * https://druginteractions.medicine.iu.edu/MainTable.aspx. Note: Please consult with the Sponsor Medical Monitor for any uncertainties regarding potential CYP3A4 and P-gp modulators.
* Active viral hepatitis, including the following:

  * Any positive test result for hepatitis B virus (HBV) indicating presence of virus, e.g., HBV DNA positive would be excluded. Participants with anti-HBs positive in line with prior vaccination or resolved infection are eligible to enroll.
  * Any positive test result for hepatitis C virus (HCV) indicating presence of active viral replication (detectable HCV RNA).
  * Participants with positive HCV antibody and an undetectable HCV RNA are eligible to enroll.
* Known human immunodeficiency virus (HIV) positive with an AIDS-defining opportunistic infection within the last year, or a current CD4 count < 350 cells/μL. Participants with HIV are eligible if they have received established antiretroviral therapy (ART) for at least 4 weeks prior to randomization and continue on ART as clinically indicated while enrolled on study. Viral serology only to be conducted if locally mandated and, if done, must be performed within 28 days of randomization.
* Evidence of active infection that requires systemic antibacterial, antiviral, or antifungal therapy ≤ 7 days prior to the first dose of study intervention.
* Live/attenuated vaccine received within 30 days of first treatment. The use of inactivated seasonal influenza vaccines (e.g., Fluzone®) will be permitted on study without restriction.
* Any botanical preparation (e.g., herbal supplements or traditional Chinese medicines) intended to treat the disease under study within 4 weeks prior to treatment. The concurrent use of any botanical preparation is not permitted while on study.
* Prior organ allograft.
* History of allergy to study intervention or any of its components.
* Known central nervous system (CNS) metastases or leptomeningeal disease is exclusionary unless adequately treated and the participant is no longer on steroids or anticonvulsants.
* Participants unable to swallow oral medication or with gastrointestinal disorders that, per the treating physician's judgement, would likely to interfere with drug absorption, are excluded.
* Pregnant or breastfeeding women are excluded.
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, or multiple allergies.

Cohort 1 specific criteria:

* Radiographically detectable metastatic disease and/or locally advanced PDAC.
* Anticipated need for preoperative radiation therapy (as determined per the treating medical team: medical oncologist and/or surgical oncologist at the time of study enrollment)

Cohort 2 specific criteria:

* Radiographically detectable metastatic disease.
* Cytotoxic chemotherapy or targeted therapy within 28 days of Cycle 1 Day 1 is not permitted. Palliative radiotherapy must have been completed 14 or more days prior to Cycle 1 Day 1.
* Participants with more than one prior line of therapy are excluded.
* Clinically significant persistent toxicities (CTCAE v5.0 Grade ≥2) caused by previous cancer therapy, excluding alopecia and Grade 2 neuropathy, are not allowed.

Cohort 3 specific criteria:

* Cytotoxic chemotherapy or targeted therapy within 28 days of Cycle 1 Day 1 is not permitted. Palliative radiotherapy must have been completed 14 or more days prior to Cycle 1 Day 1.
* Participants with more than one prior line of therapy are excluded.
* Clinically significant persistent toxicities (CTCAE v5.0 Grade ≥2) caused by previous cancer therapy, excluding alopecia and Grade 2 neuropathy, are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-05-18 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Maria P Morelli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org